CLINICAL TRIAL: NCT02717143
Title: French National Observatory Tracking Viral Myocarditis: Mortality, Cardiovascular Events, Sequels on (Magnetic Resonance Imaging) MRI
Acronym: MYOCARDITIRM
Status: Completed | Type: Observational
Sponsor: French Cardiology Society (Other)
Responsible Party: Sponsor
Other Study IDs: 15677
Record Dates: First submitted 2016-03-18; First posted 2016-03-23 (Estimated); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Myocarditis; Cardiomyopathy, Dilated; Magnetic Resonance Imaging
Keywords: Acute myocarditis; Dilated cardiomyopathy; Magnetic resonance imaging
MeSH Terms: conditions — Myocarditis; Cardiomyopathy, Dilated

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Acute myocarditis: Patients with a clinical picture suggestive of acute myocarditis: increase of troponin above the threshold defined by the pathological laboratory, associated with at least one of the three following criteria:
  1. prolonged chest pain > 10 minutes,
  2. recent infectious context <7 days
  3. young subject and / or absence of cardiovascular risk factors and / or absence of significant coronary lesion
  Patients will be included after completion of MRI confirm the diagnosis. They will be followed for 3 years, every year, by the doctor who included them in the study.
  This is an observational study that does not affect the management of patients.

SUMMARY:
Acute myocarditis is a serious illness affecting a young population with a very variable course (of full recovery at the onset of dilated cardiomyopathy (DCM), or even sudden death). Very few studies have examined the predictors of death and serious cardiovascular events in acute myocarditis and have carried on numbers of restricted patients. What little data results in a lack of a precise recommendation on the management and the follow-up period of patients.

This observational study should identify serious prognostic factor for cardiovascular events in order to provide a support strategy and more appropriate monitoring of myocarditis.

DETAILED DESCRIPTION:
Patients included in the study benefit from clinical monitoring, ultrasound and MRI as planned according to the habits of the center, regardless of the study. These clinical monitoring data, ultrasound and MRI will be collected as part of the study and if necessary telephone follow-up of cardiologists contractors will be made to complete the data. No additional examination will be conducted as part of this study. The data collected especially for cardiac MRI, will be based on the current monitoring protocol in each center.

All patients included in this study have received information and signed a consent to the use of their data during hospitalization and follow-up.

As part of this study, the inclusions are planned for a period of 2 years or more to reach a recruitment of 700 patients. The tracking target is 3 years, with an annual follow-up.

Patient follow-up is made by the doctor who selected the patient. Clinical follow-up will be made at a consultation normally provided for in hospital or cardiology practice in this type of pathology.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 years and over
* Hospitalized suspect table of acute myocarditis: Eligible patients must have an increase of troponin I greater than the threshold value of the pathological laboratory of Biochemistry, associated with at least one of the three following criteria:

  1. prolonged chest pain> 10 minutes,
  2. recent infectious context <7 days
  3. subject young and / or absence of cardiovascular risk factors and / or absence of significant coronary lesions in coronary angiography if the patient had a coronary angiography.
* Having received a cardiac MRI which concluded the diagnosis of acute myocarditis according to the usual criteria of the center (Lake Louise criteria changed according to the habits of the center) There myocarditis when at least two of the following criteria are met: hyperintense T2; hyperintense Diffusion; myocardium ratio signal / peripheral muscle Gadolinium> 4; contrast enhancement after injection of gadolinium chelate in cine-steady-state free precession (SSFP); nonischemic type of signal on delayed enhancement. These anomalies are segmental topography typically subepicardial. The analysis is made of the 17 segments of the left ventricle.
* Patient was informed and has given its consent for the study

Exclusion Criteria:

* Refusal of consent
* Claustrophobia
* Formal contraindications to MRI (allergic reaction to gadolinium chelates, porters pregnancy or patients against-indicated materials listed on the site MRI Safety "www.MRIsafety.com") :

  * Incompatible heart Pacemaker and Defibrillator
  * heart valve prostheses: valves Starr
  * Metal splinters
  * Coils intra cranial, intra cerebral surgical clips, bypass valves
  * Neurological stimulators
  * Insulin Pumps
  * Orthopedic Materials: cervical fixation with cervical Halo vest or fixer
  * Body piercing not be withdrawn

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients with clinical features of acute myocarditis previously defined and who underwent cardiac MRI which concluded the diagnosis of acute myocarditis, having agreed to participate in the study and admitted in one of the participating centers.
Sampling Method: Non-Probability Sample
Enrollment: 821 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2021-08-25 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
All cause mortality at 1 year of follow-up | 1 year
Cardiovascular mortality at 1 year of follow-up | 1 year

SECONDARY OUTCOMES:
All cause mortality at 3 years of follow-up | 3 years
Incidence of cardiovascular events at 3 years of follow-up | 3 years
  Incidence of heart failure requiring hospitalization, diagnostic of DCM not posed before the episode of myocarditis, stroke, heart transplant
Incidence of sequelae of myocarditis in cardiac MRI for patients undergoing cardiac MRI in their monitoring at 3 years of follow-up | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Phalla OU, MD. PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Claire BOULETI, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Bichat, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Magnani JW, Dec GW. Myocarditis: current trends in diagnosis and treatment. Circulation. 2006 Feb 14;113(6):876-90. doi: 10.1161/CIRCULATIONAHA.105.584532. No abstract available. PMID 16476862
- [Background] Andreoletti L, Leveque N, Boulagnon C, Brasselet C, Fornes P. Viral causes of human myocarditis. Arch Cardiovasc Dis. 2009 Jun-Jul;102(6-7):559-68. doi: 10.1016/j.acvd.2009.04.010. Epub 2009 Jul 31. PMID 19664576
- [Background] Sinagra G, Maras P, D'Ambrosio A, Gregori D, Bussani R, Silvestri F, Morgera T, Pinamonti B, Salvi A, Alberti E, Di Lenarda A, Lardieri G, Klugmann S, Camerini F. [Clinical polymorphic presentation and natural history of active myocarditis: experience in 60 cases]. G Ital Cardiol. 1997 Aug;27(8):758-74. Italian. PMID 9312504
- [Background] McCarthy RE 3rd, Boehmer JP, Hruban RH, Hutchins GM, Kasper EK, Hare JM, Baughman KL. Long-term outcome of fulminant myocarditis as compared with acute (nonfulminant) myocarditis. N Engl J Med. 2000 Mar 9;342(10):690-5. doi: 10.1056/NEJM200003093421003. PMID 10706898
- [Background] Eckart RE, Scoville SL, Campbell CL, Shry EA, Stajduhar KC, Potter RN, Pearse LA, Virmani R. Sudden death in young adults: a 25-year review of autopsies in military recruits. Ann Intern Med. 2004 Dec 7;141(11):829-34. doi: 10.7326/0003-4819-141-11-200412070-00005. PMID 15583223
- [Background] Bowles NE, Ni J, Kearney DL, Pauschinger M, Schultheiss HP, McCarthy R, Hare J, Bricker JT, Bowles KR, Towbin JA. Detection of viruses in myocardial tissues by polymerase chain reaction. evidence of adenovirus as a common cause of myocarditis in children and adults. J Am Coll Cardiol. 2003 Aug 6;42(3):466-72. doi: 10.1016/s0735-1097(03)00648-x. PMID 12906974
- [Background] Friedrich MG, Sechtem U, Schulz-Menger J, Holmvang G, Alakija P, Cooper LT, White JA, Abdel-Aty H, Gutberlet M, Prasad S, Aletras A, Laissy JP, Paterson I, Filipchuk NG, Kumar A, Pauschinger M, Liu P; International Consensus Group on Cardiovascular Magnetic Resonance in Myocarditis. Cardiovascular magnetic resonance in myocarditis: A JACC White Paper. J Am Coll Cardiol. 2009 Apr 28;53(17):1475-87. doi: 10.1016/j.jacc.2009.02.007. PMID 19389557
- [Background] Potet J, Rahmouni A, Mayer J, Vignaud A, Lim P, Luciani A, Dubois-Rande JL, Kobeiter H, Deux JF. Detection of myocardial edema with low-b-value diffusion-weighted echo-planar imaging sequence in patients with acute myocarditis. Radiology. 2013 Nov;269(2):362-9. doi: 10.1148/radiology.13121811. Epub 2013 May 21. PMID 23696680
- [Background] Caforio AL, Calabrese F, Angelini A, Tona F, Vinci A, Bottaro S, Ramondo A, Carturan E, Iliceto S, Thiene G, Daliento L. A prospective study of biopsy-proven myocarditis: prognostic relevance of clinical and aetiopathogenetic features at diagnosis. Eur Heart J. 2007 Jun;28(11):1326-33. doi: 10.1093/eurheartj/ehm076. Epub 2007 May 9. PMID 17493945
- [Background] Kindermann I, Kindermann M, Kandolf R, Klingel K, Bultmann B, Muller T, Lindinger A, Bohm M. Predictors of outcome in patients with suspected myocarditis. Circulation. 2008 Aug 5;118(6):639-48. doi: 10.1161/CIRCULATIONAHA.108.769489. Epub 2008 Jul 21. PMID 18645053
- [Background] Grun S, Schumm J, Greulich S, Wagner A, Schneider S, Bruder O, Kispert EM, Hill S, Ong P, Klingel K, Kandolf R, Sechtem U, Mahrholdt H. Long-term follow-up of biopsy-proven viral myocarditis: predictors of mortality and incomplete recovery. J Am Coll Cardiol. 2012 May 1;59(18):1604-15. doi: 10.1016/j.jacc.2012.01.007. Epub 2012 Feb 22. PMID 22365425
- [Background] Mahfoud F, Ukena C, Kandolf R, Kindermann M, Bohm M, Kindermann I. Blood pressure and heart rate predict outcome in patients acutely admitted with suspected myocarditis without previous heart failure. J Hypertens. 2012 Jun;30(6):1217-24. doi: 10.1097/HJH.0b013e328352b9ca. PMID 22473019
- [Background] Ukena C, Mahfoud F, Kindermann I, Kandolf R, Kindermann M, Bohm M. Prognostic electrocardiographic parameters in patients with suspected myocarditis. Eur J Heart Fail. 2011 Apr;13(4):398-405. doi: 10.1093/eurjhf/hfq229. Epub 2011 Jan 14. PMID 21239404
- [Background] Magnani JW, Danik HJ, Dec GW Jr, DiSalvo TG. Survival in biopsy-proven myocarditis: a long-term retrospective analysis of the histopathologic, clinical, and hemodynamic predictors. Am Heart J. 2006 Feb;151(2):463-70. doi: 10.1016/j.ahj.2005.03.037. PMID 16442915
- [Background] Mendes LA, Dec GW, Picard MH, Palacios IF, Newell J, Davidoff R. Right ventricular dysfunction: an independent predictor of adverse outcome in patients with myocarditis. Am Heart J. 1994 Aug;128(2):301-7. doi: 10.1016/0002-8703(94)90483-9. PMID 8037097
- [Derived] Bouleti C, Bejan-Angoulvant T, Servoz C, Carsten E, Genet T, Ternacle J, Deux JF, Puymirat E, Mousseaux E, Alos B, Garcia R, Bonnet G, Jacquier A, Lattuca B, Huttin O, Akodad M, Redheuil A, Angoulvant D, Ou P; MyocarditIRM Investigators. Contemporary Epidemiology, Management, and In-Hospital Outcomes of Acute Myocarditis: The Prospective Multicenter MyocarditIRM Study. JACC Heart Fail. 2025 Aug;13(8):102492. doi: 10.1016/j.jchf.2025.03.038. Epub 2025 Jun 13. PMID 40516214